Study Identifiers: DI SLE. Auto 2003; NCT 00278538

<u>Study Title</u>: Cyclophosphamide and Rabbit Antithymocyte Globulin (rATG)/Rituximab in Patients with Systemic Lupus Erythematosus

## **Statistical Analysis**

Statistical analysis was performed by the two-tailed paired student's t-test. The effects of time on the binary outcomes for IgG and IgM ACLA were evaluated using a generalized estimating equation model in SAS v9.4.